CLINICAL TRIAL: NCT03132038
Title: A Phase II, Multicenter, Non Randomized, Open Label Study of Nivolumab In Recurrent and/or Metastatic Salivary Gland Carcinoma of the Head and Neck
Brief Title: Nivolumab in Recurrent or Metastatic Salivary Gland Carcinoma of the Head and Neck
Acronym: NISCAHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0130/1619; 2016-001794-32 (EudraCT Number)
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Salivary Gland Carcinoma; Metastatic Cancer; Recurrent Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab will be given every two weeks for a maximum of one year (12 cycles) at a dose of 3 mg/kg to be administered as a 60 minute IV infusion
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg, every two weeks, during a maximum of one year
  Other Names: Opdivo

SUMMARY:
INDICATION:

Patients with recurrent and/or metastatic salivary glands carcinoma who have progressed during the 6 months period before entering the study and who are eligible for nivolumab monotherapy.

DETAILED DESCRIPTION:
METHODOLOGY:

The present study is a multicenter, open-label, non-controlled, phase II study in patients who are suffering from recurrent and/or metastatic Salivary Glands Carcinoma, who have progressed during the 6 months period before entering the study and who are eligible for nivolumab monotherapy.

All eligible patients will receive nivolumab treatment for a maximum of 12 cycles of treatment. 92 eligible patients will be dosed with nivolumab intravenously over 60 minutes (± 5 minutes) at 3 mg/kg every two weeks.

Each 28-day dosing period will constitute a cycle.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ≥18 years
* Histologically confirmed carcinoma of the salivary glands, recurrent or metastatic (adenoid cystic carcinoma or non-adenoid cystic carcinoma) not eligible to local treatment
* Pre-treatment tumor tissue available for central review and biomarkers analysis.
* At least one measurable lesion ≥10 mm (outside any previous irradiated field) according to RECIST v1.1 with magnetic resonance imaging (MRI) or computed tomography (CT)-scan
* Patients with confirmed disease progression at study entry. The "baseline" radiological evaluation (either MRI or CT scan) should demonstrate disease progression by RECIST 1.1 when compared to a prior disease assessment done within a 6 months period prior to screening
* Previous anti-cancer therapies must be discontinued at least 4 weeks prior to administration of study drug. Concomitant, palliative (limited-field) radiation therapy is permitted during the study, if all of the following criteria are met: (1) repeated imaging demonstrates no new sites of bone metastases ; (2) The lesion being considered for palliative radiation is not a target lesion
* Performance status Eastern Cooperative Oncology Group (ECOG) <2
* Screening laboratory values must meet the following criteria and should be obtained within 7 days prior to starting study drug: White Blood Cell (WBC) ≥2000/mm³, Neutrophils ≥1500/mm³, Platelets ≥100 000 /mm³, Hemoglobin >9.0 g/dL, Serum creatinine ≤1.5 x Upper Limit of Normal (ULN) or creatinine clearance (CrCl) ≥40 mL/min (using the Cockcroft-Gault formula), aspartate transaminase (AST) / alanine transaminase (ALT) / alkaline phosphatase (PAL) ≤3 x ULN or ≤5 x ULN when liver metastases, Total Bilirubin ≤1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin <3.0 mg/dL)
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab
* Women who are breastfeeding should discontinue nursing prior to the first dose of study drug and until 6 months after the last dose
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception)
* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses
* Patients with social insurance coverage

Exclusion Criteria:

* Stable disease
* Symptomatic / active brain metastases
* Immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalents) within 2 weeks prior to study drug administration. A 2 weeks wash-out minimum is required before starting study drug
* Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Patients with any active or suspected autoimmune disease or an history of known autoimmune disease (Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to an autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are however eligible for this trial)
* Patients having received prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* History of organ transplantation requiring long-term immunosuppressive medications
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Known history or active tuberculosis
* Any other malignancy (except for appropriately treated superficial basal cell skin cancer and surgically cured in situ cancer) unless free of disease for at least three years
* History of allergy to study drug components
* Any toxicity (other than alopecia) attributed to prior anti-cancer therapy not resolved to grade 1 (NCI CTCAE version 4) at baseline level before administration of study drug.
* Known or underlying medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or adverse events
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake (if applicable)
* Unwillingness to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study
* Individuals deprived of liberty or placed under the authority of a tutor
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment and during the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
non-progression rate | 6 months
  The proportion of patients with a complete response (CR) or a partial response (PR) or a stable disease (SD) as per RECIST 1.1 after 6 months of treatment.

SECONDARY OUTCOMES:
progression free survival (PFS) | the time from the date of first Nivolumab administration until the date of event, assessed up to 84 months.
  the time from the date of first Nivolumab administration until the date of event defined as the first progression according to RECIST 1.1, or death (by any cause in the absence of progression)
Overall survival | the time from the date of first dose until the date of death due to any cause, assessed up to 84 months.
  the time from the date of first dose until the date of death due to any cause
Objective response rate (ORR) | the time from the date of first dose until the date of the initial objectively documented tumor progression per RECIST v1.1 or the date of subsequent therapy, assessed up to 84 months
  ORR is defined as the number and percentage of patients with a Best Overall Response (BOR) of confirmed complete response (CR) or partial response (PR).
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | the time from the date of first dose until the end of treatment, assessed up to 84 months.
  incidence of all adverse events, serious adverse events, deaths and laboratory abnormalities
Quality of life questionnaire - Core 30 (QLQ-C30) | the time from the date of first dose until the end of treatment, assessed up to 84 months.
  Developed by the European Organisation for Research and Treatment of Cancer (EORTC), this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Head & Neck Cancer Module (QLQ-H&N35) | The time from the date of first dose until the end of treatment, assessed up to 84 months.
  This EORTC head & neck cancer specific questionnaire is intended to supplement the QLQ-C30.
  The head & neck cancer module is a 35-item questionnaire designed for use among a wide range of patients with head & neck cancer, varying in disease stage and treatment modality. It includes 7 multi-item scales that assess pain (4 items), swallowing (4 items), senses (2 items), speech (3 items), social eating (4 items), social contact (5 items), and sexuality (2 items). There are also 11 single items. Using a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), patients indicate the degree to which they have experienced symptoms. For all items and scales, high scores indicate more problems.
Biomarkers (central PD-L1 assessment, PD-L2, tumor-infiltrating lymphocyte (TILs)) | after 2 months of treatment and at the end of treatment, assessed up to 12 months.
  Correlations between expression of molecular targets and efficacy
Growth Tumor rate | At each disease evaluation from baseline to last imagery, assessed up to 84 months.
  The growth tumor rate will be assessed using RECIST 1.1 criteria before and under treatment for all eligible patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme FAYETTE, MD, Principal Investigator — Léon Bérard Center
Locations (11):
- France (11):
  - CHU Bordeaux, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Curie Saint Cloud, Saint-Cloud
  - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut de cancérologie Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
no individual participant data is shared

REFERENCES:
- [Derived] Fayette J, Even C, Digue L, Geoffrois L, Rolland F, Cupissol D, Guigay J, Le Tourneau C, Dillies AF, Zanetta S, Bozec L, Borel C, Couchon-Thaunat S, Costes-Martineau V, Sudaka-Bahadoran A, Jallut I, Garic F, Lardy-Cleaud A, Chabaud S. NISCAHN: a phase II trial of nivolumab in patients with salivary gland carcinoma (Unicancer ORL-08). BMJ Oncol. 2023 Oct 30;2(1):e000065. doi: 10.1136/bmjonc-2023-000065. eCollection 2023. PMID 39886516